CLINICAL TRIAL: NCT01068496
Title: Risk Factors and Biomarkers Associated With Recurrence After Excision of Primary Pterygium
Status: Terminated | Type: Observational
Why Stopped: Other and future studies on lipiview in pterygium will cover this current trial sufficiently.
Sponsor: Singapore National Eye Centre (Other Government)
Collaborators: Singapore Eye Research Institute (Other)
Responsible Party: Principal Investigator, Louis Tong, Singapore National Eye Centre, Singapore National Eye Centre
Other Study IDs: R707/57/2009
Record Dates: First submitted 2010-02-12; First posted 2010-02-15 (Estimated); Last update posted 2015-05-20 (Estimated); Status verified 2013-01

CONDITIONS: Pterygium
MeSH Terms: conditions — Pterygium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Pterygium and conjunctival tissue samples
Oversight: Data Monitoring Committee: No

SUMMARY:
This study looks at global gene expression in pterygium and found the derangement of matrix genes in particular to be a feature of pterygium. In the investigators opinion, it would be more beneficial to elicit changes in gene expression before the recurrence of pterygium and by developing a panel of biomarkers that are associated with pterygium recurrence; one would be able to predict the post surgical prognosis of patients after resection.Biomarker levels will be compared to discover a biomarker panel for prediction of recurrence.

DETAILED DESCRIPTION:
A comprehensive questionnaire will be used to evaluate the environmental, biological, physical and behavioral risk factors of associated with the recurrence after pterygium excision.

Slit lamp digital color photographs will be taken on primary and recurrent pterygium and pterygium will be graded in three levels of severity, based on relative transparency of pterygium tissue; grade 1 (transparent), grade 2 (intermediate), and grade 3 (opaque) to see whether the risk factors correlate to the morphology of the pterygium.

Tear samples will be collected before surgery using schirmers strip.Proteins in tear samples will be analyzed using the iTRAQ method.

The transcriptional differences in pterygium and conjunctival tissue samples will be analyzed using western blot, qPCR and immunohistochemistry assays.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of primary and recurrence pterygium
* Must agree to participate in this study
* Must sign informed consent form

Exclusion Criteria:

* Hepatitis
* HIV/AIDS

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pterygium patients from the investigator's clinic as well as other clinics at the Singapore National Eye Center will be recruited for this study.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2010-03; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
biomarkers | 12 months
  Elevation of biomarkers in pterygium tissue and tears (transcripts, proteins, or tear proteins) at the time of initial presentation of primary pterygium may predict the post-surgical recurrence within one year.
  visits: 2 further visits at 6 months and 12 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Samanthila Waduthantri, Study Chair — Singapore National Eye Centre; Laurence Lim, MBBS, Study Chair — Singapore National Eye Centre; Federico Luengo Gimeno, Study Chair — Singapore National Eye Centre; Jodhbir Mehta, Study Chair — Singapore National Eye Centre
Locations (2):
- Singapore (2):
  - Singapore National Eye Centre, Singapore, Singapore
  - Singapore National Eye Center, Singapore